CLINICAL TRIAL: NCT04556799
Title: The Clinical Results of Derotational Osteotomy Based on 3D Osteotomy Template for Treatment of Recurrent Patellar Dislocation Combined With Patellofemoral Maltracking
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Jishuitan Hospital (Other)
Responsible Party: Principal Investigator, Hui Zhang, Doctor of Sports Medicine Service of Beijing Jishuitan hospital, Beijing Jishuitan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HuiZ
Record Dates: First submitted 2020-09-15; First posted 2020-09-21 (Actual); Last update posted 2020-09-21 (Actual); Status verified 2020-09

CONDITIONS: Recurrent Patellar Dislocation; Osteotomy; Patellar Maltracking
MeSH Terms: conditions — Patellar Dislocation | interventions — Surgery, Computer-Assisted

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): 3D osteotomy template for derotation osteotomy with the aid of computer-assisted simulated surgery technique
  Interventions: Procedure: computer-assisted surgery
- Control group (Experimental): traditional osteotomy technique
  Interventions: Procedure: traditional osteotomy

INTERVENTIONS:
Procedure: computer-assisted surgery — derotation osteotomy with the aid of 3D osteotomy template and computer-assisted simulated surgery
  Arms: Study group
Procedure: traditional osteotomy — traditional osteotomy without the aid of 3D osteotomy template
  Arms: Control group

SUMMARY:
For severe recurrent patellar dislocation with poor patellar maltracking, derotation osteotomy is an effective clinical treatment. However, derotation osteotomy requires very high requirements for the surgeon. It is necessary to determine the osteotomy surface, control the axis and complete internal fixation in three dimensions. The deviation of the osteotomy surface may cause deformities such as postoperative knee valgus, knee hyperextension, or restricted extension. The hypothesis of this study is to design a 3D osteotomy template for derotation osteotomy with the aid of computer-assisted simulated surgery. Compared with traditional osteotomy, it can effectively improve the treatment effect of recurrent patellar dislocation due to poor patellar maltracking. The incidence of postoperative knee valgus shortens the operation time and reduces the number of intraoperative fluoroscopy. This study intends to adopt a randomized controlled study, and the selection criteria are adolescent patients with recurrent patellar dislocation, aged >14 years, with a positive J sign. The experimental group used mimics 20.0 software to reconstruct the three-dimensional model of the patient based on the full-length images of the lower limbs in the weight-bearing position and the CT of the hip, knee and ankle before the operation. The osteotomy template was designed and 3D printing technology was used to make the osteotomy template for intraoperative osteotomy. The control group used traditional de-rotation techniques. The knee joint range of motion, patella stability, residual rate of J-sign, knee valgus angle, femoral anteversion angle, gait analysis, etc. were compared between the two groups after surgery, and the differences between the two surgical techniques were evaluated

ELIGIBILITY:
Inclusion Criteria:

* patients with recurrent patellar dislocation
* >14 years old
* positive preoperative J-sign
* agree to participate the study

Exclusion Criteria:

* Combined with other ligament injuries of knee joint
* Skin and soft tissue conditions do not permit surgery

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-10-01 (Estimated); Primary Completion 2022-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Lysholm score | 1 year postoperatively
  A function score to assess the knee function
quadriceps strength | 1 year postoperatively
  to assess the postoperative quadriceps strength using Biodex®

CONTACTS AND LOCATIONS:
Overall Officials: Hui Zhang, Principal Investigator — Sports Medicine Service, Beijing Jishuitan hospital

IPD SHARING:
Plan to Share IPD: No